CLINICAL TRIAL: NCT06090526
Title: Pancreatic Stone Protein as Indicator for Urinary Sepsis in Intensive Care Units
Brief Title: PSP as Indicator for Urinary Sepsis in ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Maamoun Ibraheem, Doctor, Ain Shams University
Other Study IDs: biomarkes in sepsis
Record Dates: First submitted 2023-09-23; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Urinary; Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Complete blood count.
  2. Liver and kidney functions.
  3. Serum electrolytes (Na and k).
  4. C-reactive protein(CRP)
  5. Procalcitonin.
  6. PSP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: . first group (case group) will include 40 patients who will be suspected to have urinary septicemia at intensive care units of Ain Shams university.
  Interventions: Diagnostic Test: pancreatic stone protein "PSP" measurement
- control group: Second group (control group) will include 40 nonhospitalized, healthy age and sex matched adults.
  Interventions: Diagnostic Test: pancreatic stone protein "PSP" measurement

INTERVENTIONS:
Diagnostic Test: pancreatic stone protein "PSP" measurement — Blood samples will be collected for biomarker (PCT, CRP, and PSP) measurements in admission and 24 hours, 72 hours from admission and patients will be followed until death or discharge from the ICU or for 30 days, whichever occurred.

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. For clinical operationalization, organ dysfunction can be represented by an increase in the Sequential Organ Failure Assessment (SOFA) score of 2 points or more, which is associated with an in-hospital mortality greater than 10%. pancreatic stone protein has been studied as biomarker of sepsis and results suggests that it has higher diagnostic performance. The main objective of this study is to identify ability of pancreatic stone protein (PSP) as a new biomarker for diagnosis of urosepsis in Intensive Care Units comparison to other biomarkers and its role as a prognostic marker for mortality

ELIGIBILITY:
Inclusion Criteria:

* Adult ill patients at the ICU aged more than 18 years old who at risk of urosepsis.
* Both males and females.

Exclusion Criteria:

* - Age less than 18 years.
* Patients with a clinical diagnosis of sepsis at admission.
* Critically ill septic patients with a diagnosis other than urosepsis.
* Critically ill patients who were diagnosed to have urosepsis outside Ain Shams university intensive care and transferred to it.
* Malignant tumor patients.
* Uremic patients undergoing dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who was admitted in intensive care units in Ain Shams University and had risk factors for urosepsis.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
PSP ability to detect urinary sepsis | measurements from admission and patients will be followed until death or discharge from or for 30 days whichever occurred the ICU
  time course of PSP serum levels above normal range 20-50ng/ml in absence or presence of infection.

SECONDARY OUTCOMES:
PSP ability to predict prognosis of sepsis in ICU. | measurements from admission and patients will be followed until death or discharge from or for 30 days whichever occurred the ICU
  value of serial serum PSP levels from admission in ICU to predict infection severity and complications.

IPD SHARING:
Plan to Share IPD: No